CLINICAL TRIAL: NCT02301468
Title: Ischemic Compression Compared With Dry Needling as a Treatment of Myofascial Trigger Points in the Neck Region in Office Workers.
Brief Title: Ischemic Compression Compared With Dry Needling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013/903
Record Dates: First submitted 2014-11-19; First posted 2014-11-26 (Estimated); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Neck Pain; Shoulder Pain
MeSH Terms: conditions — Neck Pain; Shoulder Pain | interventions — Dry Needling; Acupressure

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dry needling (Experimental): Dry needling (experimental- physiotherapy intervention) - will be performed during 4 weeks (1 treatment/week) on the 4 most painful trigger points (determined/selected at the first session - see above). The same 4 trigger points will be treated during the 4 weeks. DN will be performed by locating the taut band and the trigger point. Once the trigger point is located, the overlying skin will be cleaned with alcohol. A certified and experienced therapist will penetrate the needle through the skin 10-15mm. into the TrP until the local twitch response will be obtained
  Interventions: Other: Dry Needling
- Ischemic compression (Experimental): Ischemic compression (experimental - physiotherapy intervention) will be performed during 4 weeks (1 treatment/week) on the 4 most painful trigger points (determined/selected at the first session - see above). IC will be performed by applying a pressure with a wooden stick on the 4 individually determined most painful trigger points. The duration of the pressure will be about 60s, (increase of pressure 10N/s) until the highest tolerable pressure will be reached and this pressure will be held even when the pain is decreasing during the intervention. The subject will always be treated by the same clinician.
  Interventions: Other: Ischemic Compression

INTERVENTIONS:
Other: Dry Needling — (experimental- physiotherapy intervention) - will be performed during 4 weeks (1 treatment/week) on the 4 most painful trigger points (determined/selected at the first session - see above). The same 4 trigger points will be treated during the 4 weeks. DN will be performed by locating the taut band and the trigger point. Once the trigger point is located, the overlying skin will be cleaned with alcohol. A certified and experienced therapist will penetrate the needle through the skin 10-15mm. into the TrP until the local twitch response will be obtained.
  Arms: Dry needling
Other: Ischemic Compression — (experimental - physiotherapy intervention) will be performed during 4 weeks (1 treatment/week) on the 4 most painful trigger points (determined/selected at the first session - see above). IC will be performed by applying a pressure with a wooden stick on the 4 individually determined most painful trigger points. The duration of the pressure will be about 60s, (increase of pressure 10N/s) until the highest tolerable pressure will be reached and this pressure will be held even when the pain is decreasing during the intervention. The subject will always be treated by the same clinician.
  Arms: Ischemic compression

SUMMARY:
A randomized controlled trial will be conducted to examine the effectiveness of DN versus IC on trigger points in the neck and shoulder region for reducing pain and improving functionality (primary outcome measures) and to investigate the effectiveness of DN versus IC for muscle strength, mobility and muscle tone (secondary outcome measures).

DETAILED DESCRIPTION:
Neck-shoulder pain is common in office workers and is characterized by pain and fatigue in this shoulder and neck region. Usually, the muscles around the neck and shoulder are involved in work-related neck-shoulder pain ( M. Trapezius, M. Levator Scapulae, M. Splenius Cervicis, M. Infraspinatus). Typically, sensitive spots are often present in the muscles, which are defined as trigger points.

In the treatment of trigger points both dry needling (DN) technique and ischemic compression (IC) technique are often used, supported by increasing scientific evidence.

In the dry needling (DN) technique a thin (acupuncture) needle punctures directly a trigger point with the aim to generate a "local twitch response". These are involuntary contractions of the muscle fibers that cause muscle relaxation and will recover the metabolism of the muscle. In the ischemic compression (IC) technique, pressure is applied slowly and progressively over the trigger point (upon the skin).

A randomized controlled trial will be conducted to examine the effectiveness of DN versus IC on trigger points in the neck and shoulder region for reducing pain and improving functionality (primary outcome measures) and to investigate the effectiveness of DN versus IC for muscle strength, mobility and muscle tone (secondary outcome measures).

To comply with these scientific objectives, 60 people will be recruited. The participants will be recruited within several business companies. The participants are people who perform at least 4 hours a day office work for at least one full year. All participants will get information and an informed consent with information about the study.

The subjects will be randomly assigned into two groups: one group treatment with DN, another group treatment with IC.

All participants are subjected to the baseline assessment. The baseline assessment includes the assessment of pain, functionality, muscle strength, mobility and muscle tone. Twelve triggerpoints (at a fixed location) will be localized and pain assessment of those trigger points will be performed. The four most painful trigger points (points at which they can tolerate the least pressure) will be determined. The treatment of both DN and IC will be performed on those 4 most painful trigger points and will last for four weeks in total (with a frequency of one treatment/week).

Two follow-up assessments will take place. A first follow-up assessment is provided one week post-intervention (short-term effects), in which all the tests are performed again. A second follow-up assessment is done at 3 months post-intervention (long-term effects).

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 18 and 65 years.
* Office workers working full time and performing at least 4 hours of computer work daily participated in this study
* >15 on the Neck Disability Index (=NDI)
* Neck-shoulder pain related to trigger points

Exclusion Criteria:

* Following treatments for their complaints
* Systemic diseases
* Neurological symptoms
* Traumatic origin of the complaints
* Pregnancy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in functionality assessment NDI (Neck Disability Index) & SPADI (Shoulder Pain and Disability Index) | at baseline, one week after the end of the treatment sessions, at 3 months
  Questionnaires : NDI (Neck Disability Index) & SPADI (Shoulder Pain and Disability Index)
Pain assessment 0-10 | at baseline
  for 12 locations of trigger points (bilaterally for Upper Trapezius , Middle Trapezius; Splenius Cervicis , Levator Scapulae , Infraspinatus, Supraspinatus ) 12 locations of trigger points will be subject to pressure of 50N. For each point, the subject will have to rate the pain on a 0-10 Numeric Rating Scale (NRS) (ranging from 0 (no pain) to 10 (worst possible pain). Based on this rating, the 4 most painful points were selected for further evaluation.
Change in Pain assessment | at baseline, one week after the end of the treatment sessions, at 3 months
  Numeric rating scale Pressure Pain Treshold from the 4 most painful trigger points ( 4 (out of 12) trigger points with the highest NRS: see 2a.) Device: Digital Pressure Algometer (compuFET; Hoggan Health Industries, Inc, West Jordan, UT) For each of the 4 most painful trigger points, the threshold will be determined as the mean of 2 consecutive (30 s in between) measurements. The PPT is the force (N) needed to give the amount of pressure that causes a changeover from sensitivity to pain in the subject.

SECONDARY OUTCOMES:
Clinical examination of the neck and the shoulder: (no pain, little pain, much pain, Movement - no limitation, little limitation, very limited) | at baseline
  Assessing pain (no pain: -, little pain: +, much pain: ++) and movement ( no limitation: - , little limitation: +, very limitated: ++ ) Neck movements: flexion - extension - sidebending ( with and without shoulder elevation), rotation and combined movements Shoulder: flexion, abduction, internal rotation, external rotation
Change in Muscle Strength Hand Held Dynamometer (CompuFet) | at baseline, one week after the end of the treatment sessions, at 3 months
  Device: Hand Held Dynamometer (CompuFet) Strength will be measured on both sides: external rotation strength test, shoulder elevation (90° of elevation in scapular plane) strength test, head extension strength test. Each test is repeated 3 times, and the mean is calculated.
Change in Mobility | at baseline, one week after the end of the treatment sessions, at 3 months
  Device: digital inclinometer ( ACUMAR Digital Inclinometer, ACU, 360°; Lafayette Instrument Company, Lafayette, IN).
  The value for 2 trials will be recorded for each direction of movement.
  * Neck: flexion, extension, sidebending bilaterally
  * Shoulder: forward flexion, abduction, internal rotation, external rotation
Change in Muscle Tone of the Trapezius muscle (bilaterally) Device: MyotonPro ® | at baseline, one week after the end of the treatment sessions, at 3 months
  Device: MyotonPro ® Placed halfway the C7 and the posterolateral part of the acromion

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Cagnie, PhD, Principal Investigator — University Ghent

REFERENCES:
- [Derived] De Meulemeester KE, Castelein B, Coppieters I, Barbe T, Cools A, Cagnie B. Comparing Trigger Point Dry Needling and Manual Pressure Technique for the Management of Myofascial Neck/Shoulder Pain: A Randomized Clinical Trial. J Manipulative Physiol Ther. 2017 Jan;40(1):11-20. doi: 10.1016/j.jmpt.2016.10.008. PMID 28017188